CLINICAL TRIAL: NCT00525525
Title: A Phase II Study of Bevacizumab Plus Temodar and Tarceva After Radiation Therapy and Temodar in Patients With Newly Diagnosed Glioblastoma or Gliosarcoma Who Are Stable Following Radiation
Brief Title: Study of Bevacizumab Plus Temodar and Tarceva in Patients With Glioblastoma or Gliosarcoma
Acronym: AVF4120s
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Michael Prados, Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07105; NCT00535249 (obsolete NCT alias)
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; Bevacizumab; Avastin; Erlotinib; Tarceva; Temozolomide; Temodar
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Bevacizumab; Erlotinib Hydrochloride; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efficacy Group (Experimental): Patients treated with the combination of radiation plus temozolomide (75 mg/m2 daily during radiotherapy) plus bevacizumab (10 mg/kg IV every two weeks during radiotherapy) plus tarceva (dose based upon use of EIAED, either 200 mg daily or 500 mg daily; given daily); all treatment begins at the start of radiotherapy and continues until tumor progression, death or excessive toxicity
  Interventions: Drug: Bevacizumab; Drug: Tarceva; Drug: Temozolomide
- Safety Lead-in Group (Other): Fractionated radiotherapy in daily doses of 1.8-2.0 Gy delivered 5 days per week over ~6 weeks, to a total dose of 59.4 to 60 Gy.
  Adjuvant temozolomide 200 mg/m^2/d x 5 d per 28-d cycle; Erlotinib 150-200 mg/d (or 500-600 mg/d for patients on enzyme-inducing antiepileptic drugs) on a continuous basis 7 days per week; Bevacizumab 10 mg/kg every 2 weeks
  Interventions: Drug: Bevacizumab; Drug: Tarceva; Drug: Temozolomide

INTERVENTIONS:
Drug: Bevacizumab — Patients are given 10 mg/kg IV Q2 weeks.
Drug: Tarceva — Patients receive 150 mg PO daily. If patients are not experiencing intolerable toxicity, they may escalate their dose to 200 mg PO daily. If patients are experiencing intolerable toxicity, their dose will be held until the toxicity improves or resolves, then re-treated at a lower dose level, i.e. 100 mg PO daily.
  Other Names: Erlotonib
Drug: Temozolomide — Patients receive 200 mg/m2 for Days 1-5 of every 28 day cycle. Although the calendar days may be slightly altered, the patient should always receive this dose for 5 days within a treatment cycle. If the patient experiences certain toxicities specified in the protocol, Temodar will be held then given at a reduced dose, i.e. 150 mg/m2 Days 1-5.

SUMMARY:
This is a phase II study of Bevacizumab plus Temodar and Tarceva in patients with non-progressive glioblastoma or gliosarcoma. Patients must have stable disease immediately following a standard course of up-front radiotherapy and Temodar. All patients will receive Bevacizumab, Temodar and Tarceva. A total of 60 patients will be enrolled. Our hypothesis is that the combination of Bevacizumab plus Temodar and Tarceva will increase survival over that seen in historical controls who have newly diagnosed, non-progressive glioblastoma or gliosarcoma following radiotherapy plus Temodar and use Temodar alone.

DETAILED DESCRIPTION:
Patients with newly diagnosed glioblastoma or gliosarcoma are treated with standard of care radiation and temozolomide, plus the addition of Bevacizumab and Tarceva. The dose of temozolomide, Bevacizumab and radiation are the same for all patients. Tarceva dose is based upon the use of enzyme inducing anti-epileptic agents. Tarceva is given daily; Bevacizumab is given every 2 weeks; radiation is for 6 weeks, and temozolomide is given daily during radiotherapy and then in the adjuvant setting, is given on a 5-day schedule every 28 days. Patients are followed for progression and survival. The measure of response is MR scanning every 2 months. Dose adjustments are based upon the specific toxicity of the agent in question which differs for each agent (Bevacizumab, temozolomide, or Tarceva). Patients are not randomized, but assigned to an arm based on use of anti-epileptic agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven, non-progressive glioblastoma multiforme (GBM) or gliosarcoma (GS) with stable disease immediately following XRT + TMZ. All patients will receive Bevacizumab plus Tarceva and TMZ.
* Biopsy or resection must have been performed prior to RT + TMZ.
* No chemotherapy is allowed prior to starting RT + TMZ, including Gliadel Wafers.
* Patients will have started RT + TMZ prior to registration and study entry and are eligible as long as they do not have progressive disease and can start Bevacizumab + TMZ and Tarceva within 4 weeks after the completion of RT + TMZ. Patients MUST have been treated with at least 54 Gy radiotherapy (60 Gy recommended) and MUST have received Temodar concurrently with radiotherapy for eligibility for this study.
* Patients may or may not have measurable or evaluable disease on contrast MR imaging. A post-radiotherapy MRI scan must document stable disease.
* Patients must be > 18 years old and with a life expectancy > 12 weeks.
* Patients must have a Karnofsky performance status of ≥ 70.
* Patients must have adequate bone marrow function (WBC > 3,000/µl, ANC > 1,500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 mg/dl), adequate liver function (SGOT and bilirubin < 1.5 times ULN), and adequate renal function (creatinine < 1.5 mg/dL) before starting therapy. These tests must be performed within 14 days prior to initial treatment.

Exclusion Criteria:

* Patients must not have evidence of recent hemorrhage on baseline MRI of the brain, with the following exceptions: presence of hemosiderin, resolving hemorrhage changes related to surgery, presence of punctuate hemorrhage in the tumor.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to tolerate this therapy or any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have proteinuria at screening as demonstrated by either

  * Urine protein: creatinine (UPC) ratio ³ 1.0 at screening OR
  * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Patients must not have inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg) on antihypertensive medications.
* Patients must not have any prior history of hypertensive crisis or hypertensive encephalopathy.
* Patients must not have New York Heart Association Grade II or greater congestive heart failure (see Appendix E).
* Patients must not have history of myocardial infarction or unstable angina within 12 months prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Clarke JL, Molinaro AM, Phillips JJ, Butowski NA, Chang SM, Perry A, Costello JF, DeSilva AA, Rabbitt JE, Prados MD. A single-institution phase II trial of radiation, temozolomide, erlotinib, and bevacizumab for initial treatment of glioblastoma. Neuro Oncol. 2014 Jul;16(7):984-90. doi: 10.1093/neuonc/nou029. PMID 24637230

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Lead-in Group: A safety lead-in group received bevacizumab and erlotinib added to TMZ after completion of radiation to rule out unexpected toxicity of the combination of drugs.
Period: Overall Study
Arm/Group | Efficacy Group | Safety Lead-in Group
Started | 59 | 15
Completed | 59 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efficacy Group | Safety Lead-in Group | Total
Number analyzed (Participants) | 59 | 15 | 74
Age, Continuous [Median (Full Range); unit: years] | 54 [21 to 76] | 65 [41 to 74] | 58 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 3 | 32
  Male | 30 | 12 | 42
Region of Enrollment [Number; unit: participants]
  United States | 59 | 15 | 74

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined from the date of diagnosis to date of death from any cause
Time Frame: Approximately 6-24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efficacy Group
Number analyzed (Participants) | 59
months | 19.8 [17.1 to 28.6]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined from the date of diagnosis to the date that progressive disease was first observed on imaging, or the date at which nonreversible neurologic progression or permanently increased corticosteroid requirement, death from any cause, or early discontinuation of treatment. Imaging guidelines were used to evaluate progression: (i) 25% increase in the sum of products of all measurable lesions over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline; (ii) clear worsening of any assessable disease; (iii) appearance of any new lesion/site; and (iv) clear clinical worsening or failure to return for evaluation as a result of death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Approximately 6 months to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efficacy Group
Number analyzed (Participants) | 59
months | 13.5 [12.2 to 17]

3. Primary Outcome: Unexpected Toxicities During First 2 Cycles of Study Drug
Description: Unexpected severe study-related adverse events
Time Frame: Within 8 weeks of initiating study therapy
Measure: Number; unit: Events
Arm/Group | Safety Lead-in Group
Number analyzed (Participants) | 15
Events | 0

ADVERSE EVENTS:
Time Frame: Duration of study treatment (up to 24 months after initial radiation)
Arm/Group | Efficacy Group | Safety Lead-in Group
Serious Adverse Events (participants affected / at risk) | 32/59 | 7/15
Other Adverse Events (participants affected / at risk) | 53/59 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efficacy Group (N=59) | Safety Lead-in Group (N=15)
Infection (Immune system disorders) | 7 | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 2
Personality/behavioral (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 8 | 1
Cerebrovascular ischemia (Vascular disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Neuropathy (Nervous system disorders) | 0 | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 1 | 0
Confusion (Nervous system disorders) | 2 | 0
Death (General disorders) | 2 | 1
Dehydration (General disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hemorrhage (CNS) (Vascular disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0
Nausea (General disorders) | 1 | 0
Headache (General disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyponatremia (Blood and lymphatic system disorders) | 2 | 0
Speech impairment (Nervous system disorders) | 2 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 1
Vomiting (General disorders) | 0 | 1
Wound complication (non-infectious) (Skin and subcutaneous tissue disorders) | 0 | 1
Weight Loss (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efficacy Group (N=59) | Safety Lead-in Group (N=15)
Diarrhea (Gastrointestinal disorders) | 5 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 | 1
Leukocytes (Blood and lymphatic system disorders) | 11 | 2
Lymphopenia (Blood and lymphatic system disorders) | 39 | 8
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 | 2
Platelets (Blood and lymphatic system disorders) | 14 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Seizure (Nervous system disorders) | 10 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Weight loss (General disorders) | 8 | 0
Anorexia (General disorders) | 0 | 2
Cardiac troponin (Cardiac disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1 | 1
Hydrocephalus (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 | 2
Mood alteration - agitation (Nervous system disorders) | 0 | 1
Nausea (General disorders) | 1 | 1
Neuropathy (Nervous system disorders) | 0 | 4
PTT (partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 | 1
Speech impairment (dysphagia/aphagia) (Nervous system disorders) | 1 | 1
Syncope (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes